CLINICAL TRIAL: NCT02820792
Title: A Randomized Non-Crossover Study of the LMA ProtectorTM Versus Ambu Aura GainTM in Adult Patients
Brief Title: Non-Crossover Study of the LMA Protector Versus Ambu AuraGain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Schulthess_Anä_8
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Airway Morbidity
MeSH Terms: interventions — Platelet Function Tests

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- LMA ProtectorTM (Active Comparator): function tests: ease of insertion, oropharyngeal seal pressure, fiberoptic position, ease of ventilation, occult blood, gastric tube insertion
  Interventions: Procedure: function tests; Device: LMA ProtectorTM
- Ambu AuraGainTM (Active Comparator): function tests: ease of insertion, oropharyngeal seal pressure, fiberoptic position, ease of ventilation, occult blood, gastric tube insertion
  Interventions: Procedure: function tests; Device: Ambu AuraGainTM

INTERVENTIONS:
Procedure: function tests — function tests: ease of insertion, oropharyngeal seal pressure, fiberoptic position, ease of ventilation, occult blood, gastric tube insertion
Device: LMA ProtectorTM
  Arms: LMA ProtectorTM
Device: Ambu AuraGainTM
  Arms: Ambu AuraGainTM

SUMMARY:
The LMA ProtectorTM is a new extraglottic airway device which brings together features of both the LMA ProSealTM (high seal cuff, gastric access and bite block - to facilitate ventilation, airway protection and airway obstruction, respectively) and the LMA UniqueTM (single use - prevention of disease transmission). In the following randomized study the investigators test the hypothesis that ease of insertion, oropharyngeal leak pressure, fiberoptic position and ease of gastric tube placement differ between the LMA ProtectorTM and the Ambu AuraGainTM in paralyzed, anesthetized patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2
* Age 19-65 yr
* Written informed consent

Exclusion Criteria:

* Difficult airway
* Non fasted
* BMI > 35

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
oropharyngeal leak pressure | 5 min
  Oropharyngeal leak pressure was determined by closing the expiratory valve of the anesthesia breathing system and a fixed gas flow of 3 l minute-1. The airway pressure at which an equilibrium was reached was noted (maximum allowed 40 cm H2O).

SECONDARY OUTCOMES:
anatomic position | 5 min
  The anatomic position was assessed by passing a fiberoptic scope through the airway tube stopping 0,5 cm prior to the end of the tube. The airway tube view was scored using an established scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Moser, MD MBA, Principal Investigator — Schulthess Klinik
Locations (2):
- Switzerland (2):
  - Schulthess Klinik, Zurich, Canton of Zurich
  - Christian Keller MD, M.Sc., Zurich

IPD SHARING:
Plan to Share IPD: No